CLINICAL TRIAL: NCT02072226
Title: A Phase IIIB, Double-Blind, Multicenter Study to Evaluate the Efficacy and Safety of Alteplase in Patients With Mild Stroke: Rapidly Improving Symptoms and Minor Neurologic Deficits (PRISMS)
Brief Title: A Study of the Efficacy and Safety of Alteplase in Participants With Mild Stroke
Acronym: PRISMS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated due to slow enrollment.
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ML29093
Record Dates: First submitted 2014-02-24; First posted 2014-02-26 (Estimated); Results first posted 2018-07-03 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-06

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Tissue Plasminogen Activator; Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Alteplase Placebo + Aspirin (Active Comparator): Participants will receive single dose of IV alteplase placebo and aspirin orally.
  Interventions: Drug: Alteplase Placebo; Drug: Aspirin
- Alteplase + Aspirin Placebo (Experimental): Participants will receive single dose of IV alteplase and aspirin placebo orally.
  Interventions: Drug: Alteplase; Drug: Aspirin Placebo

INTERVENTIONS:
Drug: Alteplase — Single dose of alteplase will be administered at 0.9 milligrams per kilogram (mg/kg) IV (maximal dose of 90 mg).
  Other Names: Activase; RO5532960
  Arms: Alteplase + Aspirin Placebo
Drug: Alteplase Placebo — Single dose of alteplase placebo will be administered as IV injection.
  Arms: Alteplase Placebo + Aspirin
Drug: Aspirin — Single dose of aspirin will be administered at 325 mg orally.
  Arms: Alteplase Placebo + Aspirin
Drug: Aspirin Placebo — Single dose of aspirin placebo will be administered orally.
  Arms: Alteplase + Aspirin Placebo

SUMMARY:
PRISMS is a double-blind, multicenter, randomized, Phase IIIb study to evaluate the efficacy and safety of intravenous (IV) alteplase in participants with mild acute ischemic strokes that do not appear to be clearly disabling. Participants will be randomized in a 1:1 ratio to receive within 3 hours of last known well time either 1) one dose of IV alteplase and one dose of oral aspirin placebo or 2) one dose of IV alteplase placebo and one dose of oral aspirin 325 milligrams (mg).

ELIGIBILITY:
Inclusion Criteria:

* Mild ischemic stroke defined as the most recent pre-treatment NIHSS score of less than or equal to(</=) 5 and determined as not clearly disabling by the investigator
* Study treatment initiated within 3 hours of last time participant seen normal

Exclusion Criteria:

* Computed tomography (CT) or magnetic resonance imaging (MRI) findings of one of the following:

  1. CT with clear large hypodensity that is greater than (>) one-third middle cerebral artery (MCA) territory (or >100 cubic centimeter [cc] if not in MCA territory)
  2. MRI with clear large hyperintensity on concurrent diffusion-weighted (DW) and fluid-attenuated inversion recovery (FLAIR) that is greater than one-third MCA territory (or greater than 100 cc if not in MCA territory),
  3. Imaging lesion consistent with acute hemorrhage, or
  4. Evidence of intraparenchymal tumor
* Disability prior to the presenting stroke
* Standard contraindications to IV alteplase within 3 hours of symptom onset, including:

  1. Head trauma, myocardial infarction, or previous stroke within the previous 3 months
  2. Gastrointestinal or urinary tract hemorrhage within the previous 21 days
  3. Major surgery within the previous 14 days
  4. Arterial puncture at non-compressible site within the previous 7 days
  5. Any history of ICH with the exception of those less than (<) 5 chronic microbleeds on MRI
  6. Elevated blood pressure defined by systolic blood pressure >185 millimeters of mercury (mm Hg) or diastolic blood pressure >110 mm Hg, or treatments requiring aggressive measures to achieve acceptable levels
  7. Treatment with unfractioned heparin within past 48 hours and activated partial thromboplastin time outside normal range
  8. Blood glucose <50 milligrams per deciliter (mg/dL)
  9. International normalized ratio >1.7
  10. Platelet count <100,000 per cubic millimeter (/mm^3)
  11. Treatment with a direct thrombin inhibitor (dabigatran) or a factor Xa inhibitor (apixaban, rivaroxaban, edoxaban) within the last 48 hours
* Allergic reaction to study drug, aspirin, or nonsteroidal anti-inflammatory drugs (NSAIDs)
* Females of childbearing age who are known to be pregnant and/or lactating
* Inability to swallow, which would prevent oral intake of aspirin or aspirin placebo tablet
* Other serious, advanced, or terminal illness that would confound the clinical outcome at 90 days
* Current or recent (within 3 months) participation in another investigational drug treatment protocol
* Anticipated inability to obtain 3-month follow-up assessments
* Previous enrollment in PRISMS
* Any other condition deemed by the investigator that would pose hazard to the participant with alteplase treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2014-05-31 (Actual); Primary Completion 2017-03-22 (Actual); Study Completion 2017-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (88):
- United States (88):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Banner Good Samaritan Medical Center, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - St. Jude Medical Center, Fullerton, California
  - University of California San Diego, La Jolla, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Hoag Memorial Hospital, Newport Beach, California
  - University of California Los Angeles, Santa Monica, California
  - Colorado Neurological Institute, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Medical Center of The Rockies, Loveland, Colorado
  - Associated Neurologists PC, Danbury, Connecticut
  - Associated Neurologists of Southern CT PC, Fairfield, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Christiana Care Health Services; Sponsor Programs Ammon Education Center, Newark, Delaware
  - Nova Clinical Research, LLC, Bradenton, Florida
  - Neurologic Consultants, P.A., Fort Lauderdale, Florida
  - University of Miami Miller School of Medicine; Clinical Reseach Building, Miami, Florida
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Alexian Brothers Neuroscience Institute, Elk Grove Village, Illinois
  - Parkview Research Center, Fort Wayne, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - St. Elizabeth Edgewood; Cancer Care Center" for Account St. Elizabeth Edgewood, Edgewood, Kentucky
  - University of Louisville, Elizabethtown, Kentucky
  - St. Elizabeth Florence, Florence, Kentucky
  - St. Elizabeth Fort Thomas, Fort Thomas, Kentucky
  - University of Kentucky, Lexington, Kentucky
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Northwest Hospital Center, Randallstown, Maryland
  - Detroit Receiving Hospital, Detroit, Michigan
  - Sparrow Health System, Lansing, Michigan
  - St Joesph Mercy Hospital Oakland, Pontiac, Michigan
  - Beaumont Hospital, Royal Oak, Michigan
  - The Minneapolis Clinic of Neurology, Golden Valley, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri Health Care, Columbia, Missouri
  - Washington University, St Louis, Missouri
  - Renown Health; Renown Institute for Neurosciences, Reno, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Shore Neurology, Toms River, New Jersey
  - SUNY Downstate Medical Center., Brooklyn, New York
  - Lutheran Medical Center, Brooklyn, New York
  - Buffalo General Medical Center, Buffalo, New York
  - Ichan School of Medicine at Mount Sinai, New York, New York
  - Columbia University Medical Center, New York, New York
  - University of North Carolina At Chapel Hill, Chapel Hill, North Carolina
  - Guilford Neurologic Associates, Greensboro, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Akron General Medical Center, Akron, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - West Hospital, Cincinnati, Ohio
  - The Christ Hospital, Cincinnati, Ohio
  - Jewish Hospital, Cincinnati, Ohio
  - Anderson Hospital, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Wright State University, Dayton, Ohio
  - Fairfield Hospital, Fairfield, Ohio
  - University of Toledo Medical Center, Toledo, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent's Medical Center, Portland, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Albert Einstein Healthcare Network, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Medical University of South Carolina; MSC 300, Charleston, South Carolina
  - University of South Carolina School of Medicine, Columbia, South Carolina
  - The Neurology And Pain Clinic, Orangeburg, South Carolina
  - Chattanooga Center for Neurologic Research, Chattanooga, Tennessee
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Valley Baptist Medical Center, Harlingen, Texas
  - Methodist Neurological Institute, Houston, Texas
  - University Of Texas Health Science Center Houston, Houston, Texas
  - Texas Tech Univ Health Sci Ctr, Lubbock, Texas
  - University Hospital San Antonio, San Antonio, Texas
  - University Of Utah, Salt Lake City, Utah
  - Inova Fairfax Hospital, Fairfax, Virginia
  - Swedish Medical Center, Seattle, Washington
  - West Virginia University Hospital, Morgantown, West Virginia
  - Gunderson Health System, La Crosse, Wisconsin
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- [Derived] Khatri P, Kleindorfer DO, Devlin T, Sawyer RN Jr, Starr M, Mejilla J, Broderick J, Chatterjee A, Jauch EC, Levine SR, Romano JG, Saver JL, Vagal A, Purdon B, Devenport J, Pavlov A, Yeatts SD; PRISMS Investigators. Effect of Alteplase vs Aspirin on Functional Outcome for Patients With Acute Ischemic Stroke and Minor Nondisabling Neurologic Deficits: The PRISMS Randomized Clinical Trial. JAMA. 2018 Jul 10;320(2):156-166. doi: 10.1001/jama.2018.8496. PMID 29998337
- [Derived] Zhao W, Mu Y, Tayama D, Yeatts SD. Comparison of statistical and operational properties of subject randomization procedures for large multicenter clinical trial treating medical emergencies. Contemp Clin Trials. 2015 Mar;41:211-8. doi: 10.1016/j.cct.2015.01.013. Epub 2015 Jan 29. PMID 25638754
- [Derived] Choi JC, Jang MU, Kang K, Park JM, Ko Y, Lee SJ, Cha JK, Kim DH, Park SS, Park TH, Lee KB, Lee J, Kim JT, Cho KH, Yu KH, Oh MS, Lee BC, Cho YJ, Kim DE, Lee JS, Lee J, Gorelick PB, Bae HJ. Comparative effectiveness of standard care with IV thrombolysis versus without IV thrombolysis for mild ischemic stroke. J Am Heart Assoc. 2015 Jan 27;4(1):e001306. doi: 10.1161/JAHA.114.000596. PMID 25628404

RESULTS

PARTICIPANT FLOW:
Groups:
- Alteplase + Aspirin Placebo: Participants received single dose of 0.9 milligram per kilogram (mg/kg) (maximal dose of 90 mg) intravenous (IV) alteplase and aspirin placebo orally.
- Alteplase Placebo + Aspirin: Participants received single dose of IV alteplase placebo and 325 mg aspirin orally.
Period: Overall Study
Arm/Group | Alteplase + Aspirin Placebo | Alteplase Placebo + Aspirin
Started | 156 | 157
Completed | 141 | 147
Not Completed | 15 | 10
Not completed — Lost to Follow-up | 11 | 7
Not completed — Patient Non-compliance | 2 | 3
Not completed — Death | 1 | 0
Not completed — Patient Withdrawal of Consent | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population included all randomized participants.
Groups:
- Alteplase + Aspirin Placebo: Participants received single dose of 0.9 mg/kg (maximal dose of 90 mg) IV alteplase and aspirin placebo orally.
- Total: Total of all reporting groups
Arm/Group | Alteplase + Aspirin Placebo | Alteplase Placebo + Aspirin | Total
Number analyzed (Participants) | 156 | 157 | 313
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.94 (13.53) | 61.20 (13.05) | 61.57 (13.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 65 | 144
  Male | 77 | 92 | 169
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 18 | 32
  Not Hispanic or Latino | 138 | 135 | 273
  Not Reported | 4 | 3 | 7
  Unknown | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 4
  Asian | 0 | 1 | 1
  Black or African American | 35 | 27 | 62
  White | 117 | 126 | 243
  Other | 1 | 0 | 1
  Unknown | 2 | 0 | 2
Total National Institutes of Health Stroke Scale (NIHSS) [Mean (Standard Deviation); unit: units on a scale] — NIHSS measures stroke symptoms. It has 11 main items which score between 0 and 4. A score of 0 typically indicates normal function, and a higher score indicates more symptoms. The individual scores from each item are summed to calculate total NIHSS score. Total NIHSS score ranges from 0 to 42, with 0 indicating no stroke symptoms, and a higher score indicating more symptoms.
  units on a scale | 2.3 (1.21) | 2.1 (1.15) | 2.2 (1.18)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Modified Rankin Scale (mRS) Score of 0 or 1 at Day 90
Description: mRS score was determined by the investigator. The mRS is a 7 point scale (0-6) with 0: No symptoms at all, 1: No significant disability despite symptoms, able to carry out all usual duties and activities, 2: Slight disability, unable to carry out all previous activities but able to look after own affairs without assistance, 3: Moderate disability requiring some help, but able to walk without assistance, 4: Moderately severe disability, unable to walk without assistance and unable to attend to own bodily needs without assistance, 5: Severe disability, bedridden, incontinent and requiring constant nursing care and attention, 6: death prior to Day 90. Reported is the percentage of participants with scores of 0 or 1 on the mRS.
Time Frame: Day 90
Population: Intent-to-Treat (ITT) population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Alteplase + Aspirin Placebo | Alteplase Placebo + Aspirin
Number analyzed (Participants) | 156 | 157
percentage of participants | 78.2 | 81.5
Statistical Analysis 1: Comparison: Alteplase + Aspirin Placebo vs Alteplase Placebo + Aspirin; Test type: Other — Confidence Interval; Adjusted Risk Difference = -1.10, 95% CI 2-sided [-9.44 to 7.25]

2. Secondary Outcome: Distribution of Participants Across the Ordinal mRS
Description: mRS score was determined by the investigator. The mRS is a 7 point scale (0-6) with 0: No symptoms at all, 1: No significant disability despite symptoms, able to carry out all usual duties and activities, 2: Slight disability, unable to carry out all previous activities but able to look after own affairs without assistance, 3: Moderate disability requiring some help, but able to walk without assistance, 4: Moderately severe disability, unable to walk without assistance and unable to attend to own bodily needs without assistance, 5: Severe disability, bedridden, incontinent and requiring constant nursing care and attention, 6: death before Day 90. Reported are the percentages of participants for all scores on the mRS.
Time Frame: Day 90
Population: ITT population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Alteplase + Aspirin Placebo | Alteplase Placebo + Aspirin
Number analyzed (Participants) | 156 | 157
percentage of participants
  mRS at Day 90 - 0 | 44.9 | 50.3
  mRS at Day 90 - 1 | 33.3 | 31.2
  mRS at Day 90 - 2 | 11.5 | 11.5
  mRS at Day 90 - 3 | 2.6 | 3.2
  mRS at Day 90 - 4 | 5.1 | 2.5
  mRS at Day 90 - 5 or 6 (death) | 2.6 | 1.3
Statistical Analysis 1: Comparison: Alteplase + Aspirin Placebo vs Alteplase Placebo + Aspirin; Test type: Other — Confidence Interval; Odds Ratio (OR) = 0.810, 95% CI 2-sided [0.527 to 1.244]

3. Secondary Outcome: Percentage of Participants With Global Favorable Recovery on mRS, NIHSS, BI, and GOS
Description: Global favorable recovery is an integrated assessment of participants who meet the following: mRS Score 0-1, National Institutes of Health Stroke Scale (NIHSS) Score 0-1, Barthel Index [BI] greater than or equal to 95, and Glasgow Outcome Scale [GOS] equal to 1. mRS Score 0-1: 0= No symptoms at all, 1= No significant disability despite symptoms, able to carry out all usual duties and activities. NIHSS Score 0-1: 0= No stroke symptoms and 1= Minor stroke symptoms. BI is a 10 question index with a total score range of 0-100 with 100 being the best outcome. GOS =1: Good recovery. Reported here are the percentages of participants who achieved a favorable score on each of these scales.
Time Frame: Day 90
Population: ITT population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Alteplase + Aspirin Placebo | Alteplase Placebo + Aspirin
Number analyzed (Participants) | 156 | 157
percentage of participants
  mRS 0 - 1 at Day 90 | 78.2 | 81.5
  NIHSS 0 - 1 at Day 90: number analyzed (Participants) | 127 | 120
  NIHSS 0 - 1 at Day 90 | 85.0 | 81.7
  BI >= 95 at Day 90: number analyzed (Participants) | 135 | 133
  BI >= 95 at Day 90 | 79.3 | 88.7
  GOS = 1 at Day 90: number analyzed (Participants) | 135 | 132
  GOS = 1 at Day 90 | 81.5 | 85.6
Statistical Analysis 1: Comparison: Alteplase + Aspirin Placebo vs Alteplase Placebo + Aspirin; Test type: Other — Confidence Interval; Odds Ratio (OR) = 0.858, 95% CI 2-sided [0.529 to 1.393]

4. Secondary Outcome: Percentage of Participants With Symptomatic Intracranial Hemorrhage (ICH )
Description: ICH was considered symptomatic if it was not seen on computed tomography (CT) or magnetic resonance imaging (MRI) scan at baseline and any neurologic decline was attributed to it by the local investigator. To detect intracranial hemorrhage, neuroimaging (CT or MRI) scan was performed at 22 to 36 hours after study drug administration.
Time Frame: Within 36 hours after study drug administration on Day 1
Population: Safety Population included all participants, who received any amount of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Alteplase + Aspirin Placebo | Alteplase Placebo + Aspirin
Number analyzed (Participants) | 154 | 153
percentage of participants | 3.2 | 0
Statistical Analysis 1: Comparison: Alteplase + Aspirin Placebo vs Alteplase Placebo + Aspirin; Test type: Other — Confidence Interval; difference in percentages = 3.25, 95% CI 2-sided [0.75 to 7.38]

5. Secondary Outcome: Percentage of Participants With Any ICH
Description: To detect ICH, neuroimaging (CT or MRI) scan was performed at 22 to 36 hours after study drug administration.
Time Frame: Within 36 hours after study drug administration on Day 1
Population: Safety Population included all participants, who received any amount of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Alteplase + Aspirin Placebo | Alteplase Placebo + Aspirin
Number analyzed (Participants) | 154 | 153
percentage of participants
  Any ICH within 36 hours reported by site | 7.1 | 2.6
  Any ICH within 36 hours reported by central reader | 7.1 | 3.3
Statistical Analysis 1: Comparison: Alteplase + Aspirin Placebo vs Alteplase Placebo + Aspirin; Any ICH within 36 hours reported by site; Test type: Other — Confidence Interval; difference in percentages = 4.53, 95% CI 2-sided [-0.34 to 10.07]
Statistical Analysis 2: Comparison: Alteplase + Aspirin Placebo vs Alteplase Placebo + Aspirin; Any ICH within 36 hours reported by central reader; Test type: Other — Confidence Interval; difference in percentages = 3.87, 95% CI 2-sided [-1.23 to 9.49]

6. Secondary Outcome: Overall Mortality
Description: Reported here is the percentage of participants who died due to any cause during the study.
Time Frame: From baseline to Day 90
Population: Safety Population included all participants, who received any amount of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Alteplase + Aspirin Placebo | Alteplase Placebo + Aspirin
Number analyzed (Participants) | 154 | 153
percentage of participants | 0.6 | 0

7. Secondary Outcome: Percentage of Participants Who Died Due to Stroke and Neurological Disorders
Description: Reported here is the percentage of participants who died due to stroke and neurological disorders.
Time Frame: From baseline to Day 90
Population: Safety Population included all participants, who received any amount of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Alteplase + Aspirin Placebo | Alteplase Placebo + Aspirin
Number analyzed (Participants) | 154 | 153
percentage of participants | 0 | 0

8. Secondary Outcome: Percentage of Participants With Adverse Events
Description: An adverse event is any untoward medical occurrence in a subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: From baseline up to Day 90: Non-serious adverse events were collected through the Day 30 visit. Serious adverse events were collected through the end of study at Day 90.
Population: Safety Population included all participants, who received any amount of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Alteplase + Aspirin Placebo | Alteplase Placebo + Aspirin
Number analyzed (Participants) | 154 | 153
percentage of participants | 77.3 | 68.0

9. Secondary Outcome: Percentage of Participants With Serious Adverse Events
Description: A serious adverse event (SAE) was defined as any experience that suggested a significant hazard, contraindication, side effect, or precaution, and fulfilled any of the following criteria: fatal (resulted in death), life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was medically significant or required intervention to prevent any of the other outcomes listed here.
Time Frame: From baseline to Day 90
Population: Safety Population included all participants, who received any amount of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Alteplase + Aspirin Placebo | Alteplase Placebo + Aspirin
Number analyzed (Participants) | 154 | 153
percentage of participants | 26.0 | 13.1

ADVERSE EVENTS:
Time Frame: Serious adverse events were collected from baseline through the end of study at Day 90. Non-serious adverse events were collected from baseline through the Day 30 visit.
Description: Safety population included all participants, who received any amount of study drug.
Arm/Group | Alteplase + Aspirin Placebo | Alteplase Placebo + Aspirin
All-Cause Mortality (participants affected / at risk) | 1/154 | 0/153
Serious Adverse Events (participants affected / at risk) | 40/154 | 20/153
Other Adverse Events (participants affected / at risk) | 49/154 | 53/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alteplase + Aspirin Placebo (N=154) | Alteplase Placebo + Aspirin (N=153)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Splenic embolism (Blood and lymphatic system disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 2 | 0
Cardiogenic shock (Cardiac disorders) | 2 | 0
Sinus node dysfunction (Cardiac disorders) | 1 | 1
Acute left ventricular failure (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Cardiac aneurysm (Cardiac disorders) | 0 | 1
Cardiac failure acute (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 1 | 0
Retinal detachment (Eye disorders) | 0 | 1
Vitreous haemorrhage (Eye disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Volvulus (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Gait disturbance (General disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Ophthalmic herpes zoster (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Fracture displacement (Injury, poisoning and procedural complications) | 1 | 0
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Haemoglobin decreased (Investigations) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 5 | 2
Stroke in evolution (Nervous system disorders) | 5 | 1
Seizure (Nervous system disorders) | 2 | 2
Transient ischaemic attack (Nervous system disorders) | 1 | 3
Haemorrhagic transformation stroke (Nervous system disorders) | 2 | 1
Carotid artery stenosis (Nervous system disorders) | 1 | 1
Cerebral haemorrhage (Nervous system disorders) | 2 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 2
Haemorrhage intracranial (Nervous system disorders) | 2 | 0
Carotid arteriosclerosis (Nervous system disorders) | 0 | 1
Embolic stroke (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 1 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Toxic encephalopathy (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 0 | 1
Device loosening (Product Issues) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Renal embolism (Renal and urinary disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alteplase + Aspirin Placebo (N=154) | Alteplase Placebo + Aspirin (N=153)
Nausea (Gastrointestinal disorders) | 9 | 13
Constipation (Gastrointestinal disorders) | 8 | 10
Hyperlipidaemia (Metabolism and nutrition disorders) | 7 | 12
Hypokalaemia (Metabolism and nutrition disorders) | 9 | 9
Headache (Nervous system disorders) | 25 | 26
Hypertension (Vascular disorders) | 11 | 10

LIMITATIONS AND CAVEATS:
The study was terminated early due to low enrollment, leading to smaller number of participants analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-05-17): https://cdn.clinicaltrials.gov/large-docs/26/NCT02072226/SAP_000.pdf
  • Study Protocol (2015-01-08): https://cdn.clinicaltrials.gov/large-docs/26/NCT02072226/Prot_001.pdf